CLINICAL TRIAL: NCT03200704
Title: Single Arm, Prospective, Open Label, Multicenter Study Assessing the Safety and Effectiveness of IC2000 and SPY Fluorescence Imaging Systems in the Visualization of Lymphatic Vessels and Lymph Nodes During Lymphatic Mapping and Sentinel Lymph Node Biopsy in Subjects With Breast Cancer
Brief Title: A Study Assessing the Safety and Effectiveness of IC2000 and SPY Fluorescence Imaging Systems (SPY-PHI) in the Visualization of Lymphatic Vessels and Identification of Lymph Nodes During Sentinel Lymph Node Biopsy in Subjects With Breast Cancer
Acronym: FILM-B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novadaq Technologies ULC, now a part of Stryker (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPY LNM 01
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Lymph Node Mapping; Sentinel Lymph Node Biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Single arm, open label, within patient study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- IC2000/SPY-PHI (Experimental): Per standard of care, each subject will receive an injection of Tc-99m radioactive colloid. Then the periareolar area of the breast(s) identified with breast cancer will be injected (intradermal) twice with 0.05 ml of a 2.5 mg/ml solution of IC2000. Following the injection lymph node mapping will occur based on intraoperative fluorescence visualization using IC2000 and SPY-PHI. Lymph nodes will be excised following identification with IC2000 and SPY-PHI. The Gamma Probe will then be used with Tc-99m for confirmation of the excised lymph nodes as well as in the area of LN excision to ensure all LNs have been identified and excised.
  Interventions: Combination Product: IC2000 and SPY-PHI; Combination Product: Tc-99m radioactive colloid and Gamma Probe

INTERVENTIONS:
Combination Product: IC2000 and SPY-PHI — Investigational treatment to assess the effectiveness of IC2000 (Indocyanine Green (ICG) for Injection) and the SPY Portable Handheld Imaging System (SPY-PHI) as an intraoperative fluorescence visualization tool, in the visual identification of lymphatic vessels and lymph nodes (LNs) during lymphatic mapping and sentinel lymph node biopsy (SLNB) procedures in early stage breast cancer
Combination Product: Tc-99m radioactive colloid and Gamma Probe — Comparator; standard of care for sentinel lymph node biopsy (SLNB) procedures in early stage breast cancer

SUMMARY:
This is a prospective, open label, multicenter, non-inferiority within-patient study to determine the effectiveness of IC2000 (Indocyanine Green (ICG) for Injection) and the SPY Portable Handheld Imaging System (SPY-PHI) as an intraoperative fluorescence visualization tool, in the visual identification of lymphatic vessels and lymph nodes (LNs) during lymphatic mapping and sentinel lymph node biopsy (SLNB) procedures as confirmed by Technitium99m (Tc99m) and Gamma Probe.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older
2. Subjects with American Cancer Society Clinical Stage 0 Ductal Carcinoma in Situ (DCIS) (Stage 0, Tis, N0, M0), IA (T1*, N0, M0), IB ((T0, N1mi, M0) or T1*, N1mi, M0)) or Stage IIA (T0, N1**M0, or T1, N1**, M0 or T2, N0, M0)1 breast cancer undergoing surgery to remove tumor draining LNs.

   Where:
   * Tis = Ductal carcinoma in situ
   * T0 = No evidence of primary tumor
   * T1 = Tumor ≤ 20 mm in greatest diameter
   * T1* = Includes T1mi
   * T2 = Tumor >20 mm but ≤ 50 mm in greatest diameter
   * N0 = No regional lymph node metastasisq1'
   * N1 = Metastasis to movable ipsilateral level I, II axillary LNs
   * N1** = T0 and T1 tumors with nodal micro-metastasis only are excluded from Stage IIA and are classified Stage IB.
   * mi = Micro-metastasis
   * M0 = Disease has not metastasized from Stage IIA and are classified Stage IB.
   * M0= No evidence of metastasis
   * mi= Micrometastasis
3. Subjects with clinically negative nodal status (N0) with or without neoadjuvant chemotherapy
4. Subjects with negative metastatic involvement (M0)
5. Subjects of child-bearing potential must not be pregnant or lactating and must have a negative pregnancy test at Baseline
6. Have signed an approved informed consent form for the study
7. Be willing to comply with the protocol

Exclusion Criteria:

1. Have had prior axillary surgery or ipsilateral radiation in the breast(s) that is planned for the procedure
2. Advanced breast cancer subjects with stage IIB, III and IV
3. Known allergy or history of adverse reaction to ICG, iodine or iodine dyes
4. Subjects who have participated in another investigational study within 30 days prior to surgery
5. Pregnant or lactating subject
6. Subjects who, in the Investigator's opinion, have any medical condition that makes the subject a poor candidate for

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Weintritt, MD, FACS, Principal Investigator — National Breast Center
Locations (7):
- United States (5):
  - Arizona Center for Cancer Care, Scottsdale, Arizona
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Methodist Dallas Medical Center, Dallas, Texas
  - Inova Health System, Alexandria, Virginia
- Canada (2):
  - Fraser Health Authority, Port Moody, British Columbia
  - CHU de Québec-Université Laval (Hôpital du Saint-Sacrement), Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects assessed for eligibility (n=153)
Period: Overall Study
Arm/Group | IC2000/SPY-PHI
Started | 152
Completed | 151
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Total enrollment (N=152)
  *PP and mITT population (N=148)
Arm/Group | IC2000/SPY-PHI
Number analyzed (Participants) | 152
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: *PP/ mITT population (N=148)
  years
    number analyzed (Participants) | 148
    (all) | 60.2 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: *PP/ mITT population (N=148)
  Participants
    number analyzed (Participants) | 148
    Female | 148
    Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: *PP/ mITT population (N=148)
  Participants
    number analyzed (Participants) | 148
    White | 120
    Black or African | 11
    Asian | 7
    Hispanic | 5
    Other | 5
Region of Enrollment [Number; unit: participants] — Population: *Please note, the region of enrollment total reflects total subjects enrolled (N=152)
  participants
    Canada | 49
    United States | 103
Smoker, n (%) [Count of Participants; unit: Participants] — Population: *PP/ mITT population (N=148)
  Participants
    number analyzed (Participants) | 148
    Current | 10
    Past | 40
    Never | 98
Alcohol consumption, n (%) [Count of Participants; unit: Participants] — Population: *PP/ mITT population (N=148)
  Participants
    number analyzed (Participants) | 148
    Yes | 75
    No | 73
Comorbid conditions of interest, n (%) [Count of Participants; unit: Participants] — Population: *PP/ mITT population (N=148)
  Participants
    number analyzed (Participants) | 148
    Hypertension | 54
    Cardiac Disease | 9
    COPD | 4
    Diabetes | 17
    Renal Failure | 2
    Liver Disease | 1
    Other | 61

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Lymph Nodes Identified by IC2000/SPY-PHI Compared to the Proportion of Lymph Nodes Identified by Tc99m/Gamma Probe
Time Frame: From Technetium-99 (Tc-99m) injection to the completion of surgery
Population: PP and mITT populations
Measure: Count of Units; unit: Lymph Nodes
Units Other Than Participants: Lymph Nodes
Arm/Group | IC2000/SPY-PHI
Number analyzed (Participants) | 148
Number analyzed (Lymph Nodes) | 406
Lymph Nodes
  Proportion of histology confirmed lymph nodes identified using IC2000 and SPY | 360
  Proportion of histology confirmed lymph nodes identified using Tc-99m/Gamma Probe | 266
Statistical Analysis 1: Comparison: IC2000/SPY-PHI; Hypothesis: H0: QT ≤ QC - 0.05 H1: QT > QC - 0.05; Test type: Non-Inferiority — 90% power, 2.5% one-sided significance level,5% non-inferiority margin; p < 0.0001, Regression, Logistic

2. Secondary Outcome: Proportion of Subjects With at Least One Lymph Node Identified by IC2000/SPY-PHI, and the Proportion of Subjects With at Least One Lymph Node Identified by Tc99m/Gamma Probe
Time Frame: From Technetium-99 (Tc-99m) injection to the completion of surgery
Population: PP and mITT population
  *The PP and mITT populations were identical
Measure: Count of Participants; unit: Participants
Arm/Group | IC2000/SPY-PHI
Number analyzed (Participants) | 148
Participants
  Proportion of Subjects with At Least One Lymph Node Identified by IC2000 and SPY in-vivo | 145
  Proportion of Subjects with At Least One Lymph Node Identified by Tc-99m/Gamma Probe | 145

3. Secondary Outcome: Proportion of Lymph Nodes Identified by IC2000/SPY-PHI by Following a Fluorescent Lymphatic Vessel, and the Proportion of Identified Lymph Nodes With no Lymphatic Vessels Visible by IC2000/SPY-PHI
Time Frame: From Technetium-99 (Tc-99m) injection to the completion of surgery
Population: Total number of histology confirmed clinical lymph nodes (specimens) identified and excised by IC2000 and SPY.
  *The PP and mITT populations were identical
Measure: Count of Units; unit: Lymph Nodes
Units Other Than Participants: Lymph Nodes
Arm/Group | IC2000/SPY-PHI
Number analyzed (Participants) | 145
Number analyzed (Lymph Nodes) | 360
Lymph Nodes
  Proportion of Lymph Nodes Identified by IC2000 and SPY in-vivo With Lymphatic Vessel Mapping | 357
  Proportion of Lymph Nodes Identified by IC2000 and SPY in-vivo Without Lymphatic Vessel Mapping | 3

4. Secondary Outcome: To Assess the Safety of Intradermal Injection of IC2000
Description: Number of subjects with treatment-related adverse events as assessed by CTCAE v5.0
Time Frame: From Technetium-99 (Tc-99m) injection to the completion of surgery
Population: Safety cohort (N=151)
Measure: Count of Participants; unit: Participants
Arm/Group | IC2000/SPY-PHI
Number analyzed (Participants) | 151
Participants | 3

ADVERSE EVENTS:
Time Frame: Collected over the treatment duration period (Day 0) and followed through to Day 30
Description: The All-Cause Mortality, Serious Adverse Event, and Adverse events are listed for the safety population and some subjects reported more than one AE or SAE.
Arm/Group | IC2000/SPY-PHI
All-Cause Mortality (participants affected / at risk) | 0/151
Serious Adverse Events (participants affected / at risk) | 4/151
Other Adverse Events (participants affected / at risk) | 27/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | IC2000/SPY-PHI (N=151)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) — A subject may have reported more than one Adverse Events.
Oxygen saturation decreased (Investigations) | 1 (1) — A subject may have reported more than one Adverse Events. *Five serious adverse events, of which one ("Apneic Episode Desaturation") was split into two different terms, 'Oxygen Saturation Decreased' and 'Apnea', therefore resulting in six SAEs.
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A subject may have reported more than one Adverse Events. *Five serious adverse events, of which one ("Apneic Episode Desaturation") was split into two different terms, 'Oxygen Saturation Decreased' and 'Apnea', therefore resulting in six SAEs.
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1/1 (1) — A subject may have reported more than one Adverse Events.
Hypertension (Vascular disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IC2000/SPY-PHI (N=151)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) — A subject may have reported more than one Adverse Events.
Angina Pectoris (Cardiac disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Atrial Fibrillation (Cardiac disorders) | 2 (2) — A subject may have reported more than one Adverse Events.
Goitre (Endocrine disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Vomiting (Gastrointestinal disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Fatigue (General disorders) | 2 (2) — A subject may have reported more than one Adverse Events.
Injection site discoloration (General disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Clostridium difficile colitis (Infections and infestations) | 1 (1) — A subject may have reported more than one Adverse Events.
Wound Infection (Infections and infestations) | 4 (4) — A subject may have reported more than one Adverse Events.
Contusion (Injury, poisoning and procedural complications) | 1 (1) — A subject may have reported more than one Adverse Events.
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1) — A subject may have reported more than one Adverse Events.
Seroma (Injury, poisoning and procedural complications) | 4 (4) — A subject may have reported more than one Adverse Events.
Skin Flap Necrosis (Injury, poisoning and procedural complications) | 1 (1) — A subject may have reported more than one Adverse Events.
Wound Secretion (Injury, poisoning and procedural complications) | 1 (1) — A subject may have reported more than one Adverse Events.
Oxygen Saturation Decreased (Investigations) | 1 (1) — A subject may have reported more than one Adverse Events.
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Chest Wall Hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Device Occlusion (Product Issues) | 2 (2) — A subject may have reported more than one Adverse Events.
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Ischemic Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Skin Discoloration (Skin and subcutaneous tissue disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Deep Vein Thrombosis (Vascular disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Flushing (Vascular disorders) | 1 (1) — A subject may have reported more than one Adverse Events.
Hypertension (Vascular disorders) | 1 (1) — A subject may have reported more than one Adverse Events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT03200704/Prot_SAP_000.pdf